CLINICAL TRIAL: NCT01100853
Title: Extended Release Naltrexone for Treating Amphetamine Dependence in Iceland
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Society of Alcoholism and other Addictions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 811095; P50DA012756 (NIH); 2009-013647-10 (EudraCT Number)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Amphetamine Dependence
Keywords: amphetamine dependence; amphetamine injection; VIVITROL/VIVITROL placebo; amphetamine craving
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended release VIVITROL injection 380 mg, 24 weeks (Active Comparator): Efficacy of 24 week course of Extended Release VIVITROL 380 mg with counseling as compared to 24 week course of VIVITROL placebo with counseling (monthly injections)
  Interventions: Drug: VIVITROL injection and VIVITROL Placebo Injection , 24 weeks
- VIVITROL placebo injection, 24 weeks (Placebo Comparator): Efficacy of 24 week course of VIVITROL with counseling as compared to 24 week course of VIVITROL placebo with counseling (monthly injections)
  Interventions: Drug: VIVITROL injection and VIVITROL Placebo Injection , 24 weeks

INTERVENTIONS:
Drug: VIVITROL injection and VIVITROL Placebo Injection , 24 weeks — Efficacy of 24 week course of VIVITROL with counseling as compared to 24 week course of VIVITROL placebo with counseling (monthly injections)

SUMMARY:
Until positive results were found with oral naltrexone, no medication has been effective against amphetamine dependence. The primary aim of this pilot study is to replicate the findings of the Swedish team that showed oral Naltrexone prevented relapse to amphetamine addiction and to extend their results by randomizing treatment-seeking amphetamine addicted patients to a 6 month course of VIVITROL (naltrexone for extended-release injectable suspension) or VIVITROL placebo. Patients in each group will receive drug counseling. VIVITROL is administered monthly and may be a better test of efficacy than tablets that must be taken daily.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above;
2. Diagnosis of amphetamine dependence as defined by DSM-IV-TR with 10 or more days of amphetamine use in the past month, and patient and clinician identify amphetamine dependence as the main problem;
3. Abstinent from substances (alcohol, amphetamines, cannabinoid, cocaine, hallucinogens, opioids, benzodiazepines [unless used to treat alcohol withdrawal] for at least 7 days prior to receiving study drug or placebo;
4. Provision of telephone numbers/contacts of three or more people that are likely to know where can be located if unable to be contacted directly;
5. Successfully complete 7-10 day assessment and study baseline measures at Vogur

Exclusion Criteria:

1. Any liver test >5 times the top limit of normal; Physiologically dependent on opioids or other substances (nicotine excepted) at time of admission to Vogur;
2. Suspected or known concomitant use of opioid analgesics, positive opioid urine drug test or positive naloxone challenge:
3. Schizophrenia, Bipolar I or other non-substance related psychotic disorder; Severely depressed, suicidal or homicidal: Dementia: Inability to understand the informed consent;
4. Planning to move from the Reykjavík area or enter jail within the next 12 months;
5. Likely to receive opioid analgesics in next 6 months associated with possible or scheduled surgery or procedure;
6. Known hypersensitivity to naltrexone, polyactide-co-glycolide (PLG); carboxymethylcellulose, or any other component of the diluent;
7. Female subjects who are pregnant or lactating, or of child bearing potential who are not using acceptable methods of birth control;
8. A body habitus that precludes use of the customized needle for intramuscular injection, based on clinical judgment;
9. Use of an investigational agent in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Pettinati, Ph.D, Principal Investigator — University of Pennsylvania; George Woody, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- SAA National Center of Addiction Medicine, Vogur Hospital, Storhofda 45, Reykjavík, Iceland

RESULTS

PARTICIPANT FLOW:
Groups:
- VIVITROL Injection, 24 Weeks; VIVITROL Placebo Injection, 24 Weeks: Efficacy of 24 week course of VIVITROL with counseling as compared to 24 week course of VIVITROL placebo with counseling (monthly injections)
Period: Overall Study
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Started | 51 | 49
Completed | 24 | 26
Not Completed | 27 | 23
Not completed — Lost to Follow-up | 11 | 6
Not completed — Received <4 study injections | 10 | 13
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 49 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.51 (1.11) | 31.59 (1.34) | 31.55 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 36 | 39 | 75
Region of Enrollment [Number; unit: participants]
  Iceland | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number Negative Urines (Proportion Negative Urines)
Time Frame: 24 Weeks
Population: Urine drug screens negative amphetamine
Measure: Number; unit: Urine Drug Screen
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Number analyzed (Participants) | 51 | 49
Urine Drug Screen | 560 | 634

2. Secondary Outcome: Amphetamine Craving Scale
Description: The Amphetamine Craving Scale is a visual analogue scale, which is scored by indicating the level of craving on a 100 mm line, where 0 is no craving at all and 100 is the highest level of craving experienced. Scores are derived from measuring their placement on the line, yielding scores from 0 to 100.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: VAS Score
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Number analyzed (Participants) | 51 | 49
VAS Score | 40.9 (4) | 46.92 (4.38)

3. Secondary Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory is a self-administered questionnaire that assess the severity of depressive symtpoms. It consists of 21 items about how the subject has been feeling in the last week, and each item has a set of at least four possible answer choices, ranging in intensity, yielding scores from 0-3, with a total possible score of 63. Higher scores indicate more severe depressive symptoms.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: BDI Score
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Number analyzed (Participants) | 51 | 49
BDI Score | 14.63 (1.40) | 14.08 (1.09)

4. Secondary Outcome: Risk Assessment Battery
Description: The Risk Assessment Battery is a 41 item self-report questionnaire that assess risk behaviors related to HIV infection over the past 6 months. The measure yields a Drug risk score ranging from 0-22 and a Sex risk score ranging from 0-18, with higher scores indicating more risk; these scores are added to yield a Total RAB score ranging from 0-40. This total scores is then divided by 40 to yield a RAB Scale Score from 0-1.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Number analyzed (Participants) | 51 | 49
Total Score | 7.14 (.62) | 5.98 (.43)

5. Secondary Outcome: Prior Admissions to Vogur Hospital
Description: Number of prior admissions due to substance dependence. The term "prior admissions" refers to admissions before enrollment, thus Baseline is the appropriate Time Frame.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of admissions
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Number analyzed (Participants) | 51 | 49
Number of admissions | 5.78 (.87) | 4.88 (.63)

6. Primary Outcome: Number Negative Urines (Proportion Negative Urines) Amphetamine
Time Frame: 24 weeks
Measure: Number; unit: Urine Drug Screen
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Number analyzed (Participants) | 51 | 49
Urine Drug Screen | 560 | 634

ADVERSE EVENTS:
Arm/Group | VIVITROL Injection, 24 Weeks | VIVITROL Placebo Injection, 24 Weeks
Serious Adverse Events (participants affected / at risk) | 9/51 | 7/49
Other Adverse Events (participants affected / at risk) | 28/51 | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIVITROL Injection, 24 Weeks (N=51) | VIVITROL Placebo Injection, 24 Weeks (N=49)
Hospitilization due to relapse to substance disorder (Psychiatric disorders) | 7 (11) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal pain, elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Potential suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIVITROL Injection, 24 Weeks (N=51) | VIVITROL Placebo Injection, 24 Weeks (N=49)
Nausea, diarrhea, discomfort/pain from stomach, heartburn (Gastrointestinal disorders) | 8 (12) | 7 (13)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (8)
Symptoms of depression and/or anxiety (Psychiatric disorders) | 5 (5) | 2 (2)
Dizziness, fatigue, fainting sensation (Nervous system disorders) | 6 (7) | 3 (3)
Elevated ALT level >5 times normal range (Hepatobiliary disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 4 (6) | 5 (6)
Other, feeling unwell, fever, loss of appetite, joint pain, pruritus, sore throat, etc. (General disorders) | 4 (9) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No